CLINICAL TRIAL: NCT05032105
Title: .An Open-label Clinical Trial Evaluating the ExAblate Model 4000 Type-1 Focused Ultrasound Unilateral Thalamotomy for Patients with Treatment-refractory Focal Onset Epilepsy and Comorbid Anxiety.
Brief Title: The Impact of Focused Ultrasound Thalamotomy of the Anterior Nucleus for Focal-Onset Epilepsy on Anxiety
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Timothy Lucas, Professor, Neurological Surgery, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023H0325
Record Dates: First submitted 2021-08-21; First posted 2021-09-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-07

CONDITIONS: Anxiety; Medication-refractory Focal-onset Epilepsy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, prospective intervention study of MRgFUSA for adults with refractory, partial-onset epilepsy with moderate-severe anxiety
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Unilateral Magnetic Resonance Imaging-guided Focused Ultrasound Ablation (MRgFUSA) of the anterior nucleus of the thalamus (ATN)
  Interventions: Device: Magnetic Resonance Imaging-guided Focused Ultrasound Ablation (MRgFUSA)

INTERVENTIONS:
Device: Magnetic Resonance Imaging-guided Focused Ultrasound Ablation (MRgFUSA) — Unilateral Magnetic Resonance Imaging-guided Focused Ultrasound Ablation (MRgFUSA) of the anterior nucleus of the thalamus (ATN)

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety, and effects on anxiety of high intensity focused ultrasound ablation (FUSA) in patients suffering from treatment-refractory focal epilepsy and anxiety. FUSA is a non-invasive neurosurgical procedure that uses ultrasound waves, sent directly through the scalp and skull, to precisely target small abnormal areas of the brain. For this study, the targeted area of the brain is the anterior nucleus of the thalamus. This brain region may cause seizures and may also be involved in anxiety. The study will test if FUSA is safe and tolerated, and if it reduces anxiety and brain response to threat in patients with anxiety receiving the procedure for partial-onset epilepsy that is resistant to medications.

DETAILED DESCRIPTION:
This is an open-label, Phase 1 prospective intervention study. Ten (10) adults with refractory, partial-onset epilepsy with moderate-severe anxiety and able to provide informed consent will be enrolled.

Patients, eligible for Magnetic Resonance Imaging-guided Focused Ultrasound Ablation (MRgFUSA) of the anterior nucleus of the thalamus (ATN) for treatment-refractory epilepsy and who present moderate-severe anxiety will be enrolled. In addition to the diagnosis of medically refractory epilepsy, patients will need to present moderate to severe anxiety (as measured by the Hamilton Anxiety Rating Scale, HAM-A; HAMA score > 17) and other protocol specific inclusion and exclusion criteria.

Medication-refractory partial or focal-onset epilepsy is often associated with enhanced fear behaviors and clinical anxiety. Exaggerated amygdala reactivity to threat is a cardinal neural phenotype of fear and anxiety disorders. The study will determine if MRgFUSA-ATN is feasible and safe and its effects on anxiety, using neuroimaging and neurological, neurocognitive/neuropsychological, psychiatric assessments before, and 1 day, 1 week, 1 month, 3 months, 6 months and 12 months post MRgFUSA.

Feasibility is defined as the ability to create the desired lesion within the anterior nucleus of the thalamus and perform fMRI to measure threat reactivity.

Safety will be measured by recording and analyzing any adverse effects that may occur from before surgery through 12 months following the surgery. These will include any new onset of neurological deficits, or performance deterioration on neuropsychological testing.

Effects on anxiety will be measured using amygdala reactivity to threat by fMRI and patient- and clinician-reported measures of anxiety symptoms before and after MRgFUSA-ATN up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Disabling, medically refractory epilepsy (≥2 anti-epileptic drug failures).
* Focal onset seizures with secondary generalization; with or without primary generalized seizures.
* Previous seizure work-up within 12 months of enrollment date to include:

A. Home EEG or EMU video EEG or intracranial EEG. B. High definition MRI imaging/PET imaging. C. Baseline neuropsychological assessment, which includes the Wechsler Advanced Clinical Solutions - Test of Premorbid Functioning (TOPF).

* ≥ 3 seizures/month on average within 3 months of enrollment.
* Stable medication (including anti-epileptic and psychotropic/psychoactive medications) dosage for 3 months before enrollment.
* Moderate-severe anxiety as measured by the Hamilton Anxiety Rating Scale (HAM-A) score > 17.
* Anterior Nucleus (AN) identifiable on MRI (structural T1 and T2 images).
* Willing to maintain seizure diary (3 months before & 3 months after).
* Involved care provider.
* Written informed consent to participate.
* Ability to comply with all testing, follow-ups, and study appointments and protocols.

Exclusion Criteria:

* Low seizure frequency (<3 seizures/month).
* Generalized epilepsy (Lennox Gastaut, drop attacks).
* Post infectious epilepsy (post herpetic).
* Unable or unwilling to maintain anti-epilepsy drug dosage for 3 months post treatment.
* Active (current in past 12 months), uncontrolled DSM-5 psychiatric disorder, except for anxiety disorders.
* Recent (past 12 months) history of drugs or alcohol abuse as evidenced by diagnosis of Substance Use Disorder.
* Active suicidal ideation current and past 30 days.
* Clinically significant neurological disorder, except for epilepsy.
* Presence of any neurodegenerative disease suspected on neurological examination. These include but are not limited to: Multisystem atrophy; Progressive supranuclear palsy; Dementia with Lewy bodies; Alzheimer's disease; Parkinson's disease.
* Cerebrovascular disease (multiple CVA or CVA within six months).
* Significant structural brain abnormalities.
* Surgical lesion identifiable on imaging.
* Symptoms and signs of increased intracranial pressure.
* Patients with any types of brain tumors, including metastases.
* Previous vagal nerve stimulator.
* Previous corpus callosotomy.
* Patients who have had deep brain stimulation.
* Prior stereotactic ablation.
* Positive urine drug screen at study entry or any follow-up testing session. For cannabis, exclusion includes positive drug screen with self-report of cannabis use in the past 48 hours.
* Known allergic reaction and/or hypersensitivity to IV dye and/or IV contrasting agent(s).
* Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* History of claustrophobia.
* Unstable cardiac status including: Unstable angina pectoris on medication; documented myocardial infarction within last 40 days to protocol entry; Congestive heart failure; Severe hypertension (diastolic BP> 100 on medication).
* Patients receiving dialysis;
* Patients with risk factors for intraoperative or postoperative bleeding: Platelet count less than 100,000 per cubic millimeter; PT> 14PTT > 40; INR > 1.43.
* History of abnormal bleeding and/or coagulopathy.
* Receiving anticoagulant (e.g., Warfarin) or antiplatelet (e.g., aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk of hemorrhage (e.g., Avastin) within one month of scheduled focused ultrasound procedure.
* History of intracranial hemorrhage.
* Active or suspected, acute or chronic uncontrolled infection or known life-threatening systemic disease;
* History of immunocompromised status, including patients who are HIV positive.
* Subjects with remarkable atrophy and poor healing capacity of the scalp.
* Evidence for calcifications that might interfere with treatment safety (per CT).
* Skull Density Ratio (SDR) <0.4.
* Pregnancy or lactation or planning to become pregnant during the time-period of the study.
* Any illness that in the investigators' opinion preclude participation in this study.
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time);
* IQ score of <70 on the Wechsler Advanced Clinical Solutions - Test of Premorbid Functioning (TOPF), measured as part of screening neuropsychological assessment.
* Presence of significant cognitive impairment as determined with a score ≤24 on the Mini Mental Status Examination (MMSE).
* Patients unable to communicate with the investigator and staff.
* Legal incapacity or limited legal capacity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
  Safety will be determined by an evaluation of the incidence and severity of MRgFUSA-ATN and other research procedures related adverse events from the 1st study visit through the 12-month post-treatment time point. Post-procedural imaging will be evaluated for evidence of swelling, hemorrhage, and the evolution of the ATN lesion. Emergence of complications will be monitored by neurological examination at day 1, day 7, month 1, month 3, month 6 and month 12 post-procedure. A comprehensive battery of neuropsychological assessments will be conducted by board-certified neuropsychologists at study screening, 3-month and 12-month postoperative time points. All events that are not procedure related will also be captured and recorded.
Target | 1 month
  Feasibility will be determined by ability to create the desired lesion within the anterior nucleus of the thalamus as assessed by neuroimaging
Change in Anxiety symptoms | 12 months
  Change in anxiety symptoms will be measured using clinician-administered HAM-A scale before the procedure and at various time points after the procedure.
  HAM-A is the scale of reference used in clinical trials to rate the severity of symptoms of anxiety in patients. It will be collected before and after the procedure at day 1, 7, months 1, 3, 6 and 12 to determine any effect and its change overtime.
Effect on Threat Reactivity | 1 day
  Change in Threat reactivity measured by fMRI task just before and after MRgFUSA

SECONDARY OUTCOMES:
Change in seizure frequency | 12 months
  Change in seizure frequency between before the procedure and after will be assessed by online or hard copy seizure diary
Ability to perform the threat reactivity fMRI task just before and after MRgFUSA | 4 years
  Ability to perform the fMRI task before and after MRgFUSA will be assessed by recording any delay or inability to perform the assessment
Change in self-reported anxiety symptoms | 12 months
  Change in Self-report symptoms of anxiety using the Beck Anxiety Inventory from before the procedure up to 12 months post-procedure.
Change in self-reported anxiety symptoms | 12 months
  Change in Self-report symptoms on the Anxiety, Depression, Stress scale from before the procedure up to 12 months post-procedure
Change in quality of life | 12 months
  Change in quality of life between before and after the procedure will be measured using the Quality of Life in Epilepsy Inventory before and up to 12 months after the procedure
Rate of Patient Accrual | 4 years
  Feasibility will be assessed by measuring the rate of patient accrual over the 4 years of the study

CONTACTS AND LOCATIONS:
Overall Officials: Kinh Luan Phan, MD, Principal Investigator — Ohio State University; Timothy Lucas, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared via the NIMH Data Archive, in compliance with NIH policy

REFERENCES:
- [Background] Rabut C, Yoo S, Hurt RC, Jin Z, Li H, Guo H, Ling B, Shapiro MG. Ultrasound Technologies for Imaging and Modulating Neural Activity. Neuron. 2020 Oct 14;108(1):93-110. doi: 10.1016/j.neuron.2020.09.003. PMID 33058769
- [Background] Krishna V, Sammartino F, Rezai A. A Review of the Current Therapies, Challenges, and Future Directions of Transcranial Focused Ultrasound Technology: Advances in Diagnosis and Treatment. JAMA Neurol. 2018 Feb 1;75(2):246-254. doi: 10.1001/jamaneurol.2017.3129. PMID 29228074
- [Background] Kim M, Kim CH, Jung HH, Kim SJ, Chang JW. Treatment of Major Depressive Disorder via Magnetic Resonance-Guided Focused Ultrasound Surgery. Biol Psychiatry. 2018 Jan 1;83(1):e17-e18. doi: 10.1016/j.biopsych.2017.05.008. Epub 2017 May 12. No abstract available. PMID 28601192
- [Background] Jung HH, Kim SJ, Roh D, Chang JG, Chang WS, Kweon EJ, Kim CH, Chang JW. Bilateral thermal capsulotomy with MR-guided focused ultrasound for patients with treatment-refractory obsessive-compulsive disorder: a proof-of-concept study. Mol Psychiatry. 2015 Oct;20(10):1205-11. doi: 10.1038/mp.2014.154. Epub 2014 Nov 25. PMID 25421403
- [Background] Davidson B, Hamani C, Rabin JS, Goubran M, Meng Y, Huang Y, Baskaran A, Sharma S, Ozzoude M, Richter MA, Levitt A, Giacobbe P, Hynynen K, Lipsman N. Magnetic resonance-guided focused ultrasound capsulotomy for refractory obsessive compulsive disorder and major depressive disorder: clinical and imaging results from two phase I trials. Mol Psychiatry. 2020 Sep;25(9):1946-1957. doi: 10.1038/s41380-020-0737-1. Epub 2020 May 14. PMID 32404942
- [Background] Lipsman N, Schwartz ML, Huang Y, Lee L, Sankar T, Chapman M, Hynynen K, Lozano AM. MR-guided focused ultrasound thalamotomy for essential tremor: a proof-of-concept study. Lancet Neurol. 2013 May;12(5):462-8. doi: 10.1016/S1474-4422(13)70048-6. Epub 2013 Mar 21. PMID 23523144
- [Background] Hingray C, McGonigal A, Kotwas I, Micoulaud-Franchi JA. The Relationship Between Epilepsy and Anxiety Disorders. Curr Psychiatry Rep. 2019 Apr 29;21(6):40. doi: 10.1007/s11920-019-1029-9. PMID 31037466
- [Background] Jackson MJ, Turkington D. Depression and anxiety in epilepsy. J Neurol Neurosurg Psychiatry. 2005 Mar;76 Suppl 1(Suppl 1):i45-47. doi: 10.1136/jnnp.2004.060467. No abstract available. PMID 15718221
- [Background] Janiri D, Moser DA, Doucet GE, Luber MJ, Rasgon A, Lee WH, Murrough JW, Sani G, Eickhoff SB, Frangou S. Shared Neural Phenotypes for Mood and Anxiety Disorders: A Meta-analysis of 226 Task-Related Functional Imaging Studies. JAMA Psychiatry. 2020 Feb 1;77(2):172-179. doi: 10.1001/jamapsychiatry.2019.3351. PMID 31664439
- [Background] Etkin A, Wager TD. Functional neuroimaging of anxiety: a meta-analysis of emotional processing in PTSD, social anxiety disorder, and specific phobia. Am J Psychiatry. 2007 Oct;164(10):1476-88. doi: 10.1176/appi.ajp.2007.07030504. PMID 17898336
- [Background] Gorka SM, Young CB, Klumpp H, Kennedy AE, Francis J, Ajilore O, Langenecker SA, Shankman SA, Craske MG, Stein MB, Phan KL. Emotion-based brain mechanisms and predictors for SSRI and CBT treatment of anxiety and depression: a randomized trial. Neuropsychopharmacology. 2019 Aug;44(9):1639-1648. doi: 10.1038/s41386-019-0407-7. Epub 2019 May 6. PMID 31060042
- [Background] Phan KL, Coccaro EF, Angstadt M, Kreger KJ, Mayberg HS, Liberzon I, Stein MB. Corticolimbic brain reactivity to social signals of threat before and after sertraline treatment in generalized social phobia. Biol Psychiatry. 2013 Feb 15;73(4):329-36. doi: 10.1016/j.biopsych.2012.10.003. Epub 2012 Nov 17. PMID 23164370
- [Background] Sripada CS, Angstadt M, McNamara P, King AC, Phan KL. Effects of alcohol on brain responses to social signals of threat in humans. Neuroimage. 2011 Mar 1;55(1):371-80. doi: 10.1016/j.neuroimage.2010.11.062. Epub 2010 Nov 29. PMID 21122818
- [Background] Paulus MP, Feinstein JS, Castillo G, Simmons AN, Stein MB. Dose-dependent decrease of activation in bilateral amygdala and insula by lorazepam during emotion processing. Arch Gen Psychiatry. 2005 Mar;62(3):282-8. doi: 10.1001/archpsyc.62.3.282. PMID 15753241
- [Background] Salanova V, Witt T, Worth R, Henry TR, Gross RE, Nazzaro JM, Labar D, Sperling MR, Sharan A, Sandok E, Handforth A, Stern JM, Chung S, Henderson JM, French J, Baltuch G, Rosenfeld WE, Garcia P, Barbaro NM, Fountain NB, Elias WJ, Goodman RR, Pollard JR, Troster AI, Irwin CP, Lambrecht K, Graves N, Fisher R; SANTE Study Group. Long-term efficacy and safety of thalamic stimulation for drug-resistant partial epilepsy. Neurology. 2015 Mar 10;84(10):1017-25. doi: 10.1212/WNL.0000000000001334. Epub 2015 Feb 6. PMID 25663221
- [Background] Ranjan M, Boutet A, Bhatia S, Wilfong A, Hader W, Lee MR, Rezai AR, Adelson PD. Neuromodulation beyond neurostimulation for epilepsy: scope for focused ultrasound. Expert Rev Neurother. 2019 Oct;19(10):937-943. doi: 10.1080/14737175.2019.1635013. Epub 2019 Jul 2. PMID 31232614
- [Background] So RQ, Krishna V, King NKK, Yang H, Zhang Z, Sammartino F, Lozano AM, Wennberg RA, Guan C. Prediction and detection of seizures from simultaneous thalamic and scalp electroencephalography recordings. J Neurosurg. 2017 Jun;126(6):2036-2044. doi: 10.3171/2016.7.JNS161282. Epub 2016 Oct 7. PMID 27715438
- [Background] Biraben A, Taussig D, Thomas P, Even C, Vignal JP, Scarabin JM, Chauvel P. Fear as the main feature of epileptic seizures. J Neurol Neurosurg Psychiatry. 2001 Feb;70(2):186-91. doi: 10.1136/jnnp.70.2.186. PMID 11160466
- [Background] Krishna V, Sammartino F, Cosgrove R, Ghanouni P, Schwartz M, Gwinn R, Eisenberg H, Fishman P, Chang JW, Taira T, Kaplitt M, Rezai A, Rumia J, Gedroyc W, Igase K, Kishima H, Yamada K, Ohnishi H, Halpern C. Predictors of Outcomes After Focused Ultrasound Thalamotomy. Neurosurgery. 2020 Aug 1;87(2):229-237. doi: 10.1093/neuros/nyz417. PMID 31690945
- [Background] Boulogne S, Catenoix H, Ryvlin P, Rheims S. Long-lasting seizure-related anxiety in patients with temporal lobe epilepsy and comorbid psychiatric disorders. Epileptic Disord. 2015 Sep;17(3):340-4. doi: 10.1684/epd.2015.0757. PMID 26235301
- [Background] Krishna V, King NK, Sammartino F, Strauss I, Andrade DM, Wennberg RA, Lozano AM. Anterior Nucleus Deep Brain Stimulation for Refractory Epilepsy: Insights Into Patterns of Seizure Control and Efficacious Target. Neurosurgery. 2016 Jun;78(6):802-11. doi: 10.1227/NEU.0000000000001197. PMID 26813858
- [Background] Sammartino F, Yeh FC, Krishna V. Longitudinal analysis of structural changes following unilateral focused ultrasound thalamotomy. Neuroimage Clin. 2019;22:101754. doi: 10.1016/j.nicl.2019.101754. Epub 2019 Mar 12. PMID 30921612